CLINICAL TRIAL: NCT02329561
Title: Comparative, Randomized, Double-Blind, Single-Dose, 2-way Crossover Study to Evaluate the Pharmacokinetics and Analgesic Effect of Labopharm Tramadol Contramid® OAD 200 mg Tablets or Placebo in Healthy Young and Elderly Adult Volunteers
Brief Title: PK PD of the Enantiomers of Tramadol and O-desmethyltramadol in Elderly and Young Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Labopharm Inc. (Industry); MDS Pharma Services (Industry)
Responsible Party: Principal Investigator, France Varin, France Varin B. Pharm. Ph.D, Full Professer, Université de Montréal
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MDT1-20
Record Dates: First submitted 2014-12-19; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Aging; Pain
Keywords: Pharmacokinetics; Opioid; Geriatric; Pharmacodynamics
MeSH Terms: conditions — Pain | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol extended release and CP/T (Active Comparator): Tramadol extended release: 200mg Single-dose, extended-release, once-daily, tablet; Current Perception and Tolerance (CP/T)
  Interventions: Drug: Tramadol extended release 200 mg; Behavioral: CP/T
- Placebo and CP/T (Placebo Comparator): Single-dose, placebo identical in appearance to an extended release once-daily tablet; Current Perception and Tolerance (CP/T)
  Interventions: Behavioral: CP/T; Drug: Placebo

INTERVENTIONS:
Drug: Tramadol extended release 200 mg — Tramadol extended release 200 mg: Administration of a single 200mg tramadol extended-release tablet
  Other Names: Tramadol Contramid 200 mg extended-release
  Arms: Tramadol extended release and CP/T
Behavioral: CP/T — Subjects were evaluated for perception and tolerance of electrical current. An experimentally induced pain model utilizing electrical stimulation from the FDA approved Neurometer, as the painful stimulus was used to assess Current Perception Threshold and Pain Tolerance Threshold (CP/T) in young and elderly subjects following administration of tramadol and of placebo.
  Other Names: Electrically stimulated experimental pain model (ESEPM)
Drug: Placebo — Administration of a single placebo tablet identical in appearance to a 200mg tramadol extended-release tablet
  Other Names: sugar pill
  Arms: Placebo and CP/T

SUMMARY:
This study evaluates the pharmacokinetics and pharmacodynamics of the enantiomers of tramadol and O-desmethyltramadol (ODM) in generally healthy young and elderly adults. Using a randomised, double-blind, crossover design, participants were administered a single 200mg tramadol extended-release tablet and placebo.

DETAILED DESCRIPTION:
The pharmacokinetics of the enantiomers of tramadol and O-desmethyltramadol (ODM) have not been extensively studied in elderly patients. Given the importance of hepatic function in the metabolism of tramadol into the more potent ODM metabolite and the fact that tramadol is primarily renally excreted, age-related changes in hepatic and renal function may affect the pharmacokinetics and pharmacodynamics of tramadol. Data on the pharmacokinetics of tramadol, the ODM metabolite and their enantiomers will provide important information as to the source of any differences in the metabolism or elimination of Tramadol Contramid® OAD in the elderly as compared to younger subjects. Differences in the PK of tramadol and O-desmethyltramadol could result in differences in Pharmacodynamics of tramadol, specifically in analgesic effect. An Electrically Stimulated Pain Model was used to evaluate any differences in current perception and pain tolerance between the age groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteers, 18-40 years of age.
* Adult male or female volunteers aged 75 years or more
* Subjects with a BMI less than 35 kg/m2.
* Generally healthy, elderly subjects with mild renal impairment (creatinine clearance 50-80 mL/min or glomerular filtration rate ≥ 50 mL/min/1.73 m2) or mild hepatic impairment (Child-Pugh Class A)
* Medically stable healthy subjects with non-clinically significant laboratory profiles, vital signs and ECGs.
* Subjects will be non-smokers for at least 3 months prior to the first dose or consistent moderate smokers (fewer than 10 cigarettes per day) for at least 3 months prior to the first dose.
* Females of childbearing potential must be using medically acceptable birth control methods
* Voluntary written informed consent

Exclusion Criteria:

* History or presence of significant unstable or untreated cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* alcoholism or drug abuse within the past year;
* previous or current opioid dependency or other substance abuse or dependence, other than nicotine;
* hypersensitivity or idiosyncratic reaction to tramadol hydrochloride, codeine, opioids or other synthetic opioids of the aminocyclohexanol group;
* seizures (other than infantile febrile seizures);
* significant head trauma.
* Subjects who tested positive at screening for HIV, HBsAg or HCV.
* Subjects whose sitting blood pressure is less than 110/60 mmHg at screening or prior to dosing.
* Subjects whose pulse is lower than 55 b.p.m. at screening or prior to dosing for young subjects or less than 60 b.p.m at screening or prior to dosing for the elderly subjects.
* Subjects who have used any drugs or substances known to be strong inhibitors of CYP enzymes (formerly known as cytochrome P450 enzymes) within 10 days prior to the first dose.
* Subjects who have used any drugs or substances known to be strong inducers of CYP enzymes (formerly known as cytochrome P450 enzymes) within 28 days prior to the first dose.
* Subjects who are revealed upon genotyping to be CYP2D6 poor metabolisers.
* Subjects who have received monoamine oxidase inhibitors (MAOI) or antidepressants (tricyclic or SSRIs), within 28 days prior to the first dose.
* Subjects who have received drugs belonging to the opioids/analgesic class, within 5 elimination half-lives prior to the first dose.
* Subjects who have received coumarin derivatives (e.g warfarin) or digoxin, within 28 days prior to the first dose.
* Subjects who have received CNS depressant drugs (such as benzodiazepines, barbiturates, sedative H1 antihistamines, neuroleptics, some beta-blockers, anxiolytics other than benzodiazepines), tricyclic compounds (such as cyclobenzaprine, promethazine), drugs increasing serotonin levels or thalidomide within 5 elimination half-lives prior to the first dose.
* Subjects with significant liver disease (Child-Pugh Score greater than or equal to 7).
* Significant renal disease as determined by the Cockcroft-Gault formula
* Bowel disease affecting absorption.
* Major illness requiring hospitalization during the last 3 months prior to the first dose.
* Previous failure of treatment with tramadol or discontinuation of treatment with tramadol due to adverse events.
* Subjects who have been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Subjects who have any condition that, in the opinion of the Investigator, makes the subject unsuitable for the study.
* Subjects who donated significant amounts of blood in the last year
* Subjects who have participated in another clinical trial within 28 days prior to the first dose.
* Subjects who are unable to tolerate the training for the ESEPM.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To characterise and compare the pharmacokinetic parameters of AUC 0-t, AUCinf, Cmax, tmax, t½, CL/F, Varea/F, Ae 0 48, Rmax and CLr for the enantiomers of tramadol and O-desmethyltramadol in young and elderly subjects | 48 hours
  To characterise and compare the pharmacokinetic parameters of AUC 0-t, AUCinf, Cmax, tmax, t½, CL/F, Varea/F, Ae 0 48, Rmax and CLr for the enantiomers of tramadol and O-desmethyltramadol in healthy adult young and elderly subjects. Plasma samples were taken at 16 timepoints throughout 48 hours and evaluated for plasma concentrations of (+)- and (-)- tramadol

SECONDARY OUTCOMES:
To characterise and compare threshold of current perception in young and elderly subjects | 30 hours
  Healthy adult young and elderly subjects were tested to determine the milliamperes of current that resulted in perception of an electrical stimulus in the non-dominant forefinger at 15 timepoints throughout 30 hours using an electrically stimulated pain model after treatment with active drug and placebo with random assignment of treatment sequence (placebo then tramadol or tramadol then placebo)
To characterise and compare threshold of pain tolerance in young and elderly subjects | 30 hours
  Healthy adult young and elderly subjects were tested to determine the milliamperes of current they were willing to tolerate at 15 timepoints throughout 30 hours using an electrically stimulated pain model after treatment with active drug and placebo with random assignment of treatment sequence (placebo then tramadol or tramadol then placebo)

CONTACTS AND LOCATIONS:
Overall Officials: France Varin, BPharm, PhD, Principal Investigator — Université de Montréal

REFERENCES:
- [Derived] Robertson SS, Mouksassi MS, Varin F. Population Pharmacokinetic/Pharmacodynamic Modeling of O-Desmethyltramadol in Young and Elderly Healthy Volunteers. Drugs Aging. 2019 Aug;36(8):747-758. doi: 10.1007/s40266-019-00681-w. PMID 31161580
- [Derived] Skinner-Robertson S, Fradette C, Bouchard S, Mouksassi MS, Varin F. Pharmacokinetics of Tramadol and O-Desmethyltramadol Enantiomers Following Administration of Extended-Release Tablets to Elderly and Young Subjects. Drugs Aging. 2015 Dec;32(12):1029-43. doi: 10.1007/s40266-015-0315-4. PMID 26508138